CLINICAL TRIAL: NCT05322733
Title: Efficacy and Safety of Orelabrutinib, Fludarabine, Cyclophosphamide, and Obinutuzumab (GA-101) (oFCG) in the Treatment of Newly Diagnosed Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL)
Brief Title: Orelabrutinib and Obinutuzumab Plus FC Regimen in Treating Newly Diagnosed CLL/SLL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWCLL-001
Record Dates: First submitted 2022-03-09; First posted 2022-04-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — orelabrutinib; obinutuzumab; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (oFCG) (Experimental): See Detailed Description.
  Interventions: Drug: Orelabrutinib; Drug: Obinutuzumab; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Orelabrutinib — 150 mg capsules administered orally once daily (28-day cycles). Until 12 or 24 cycles and following BM undetectable MRD, or disease progression, or intolerant toxicity.
  Other Names: ICP-022
Drug: Obinutuzumab — 1000 mg administered intravenously once on Day 1, 8, 15 of first cycle and on Day 1 of following cycles for maximal 12 cycles (28-day cycles).
  Other Names: GA101
Drug: Fludarabine — 25mg/m2/day administered intravenously on Day 1-3 for every cycle (at most 6 cycles, 28-day cycles).
  Other Names: Fludara
Drug: Cyclophosphamide — 250mg/m2/day administered intravenously on Day 1-3 for every cycle (at most 6 cycles, 28-day cycles).

SUMMARY:
This study is a multi-center, open-label, single-arm, non-randomized phase II clinical study in order to evaluate the safety and efficacy of Orelabrutinib, Fludarabine, Cyclophosphamide, and Obinutuzumab (GA-101) (oFCG) in the Treatment of Newly Diagnosed Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL)

DETAILED DESCRIPTION:
Patients eligible for enrollment will receive 7-day lead-in therapy of orelabrutinib 150 mg once daily, followed by 3 cycles of orelabrutinib, fludarabine, cyclophosphamide, and obinutuzumab (oFCG) at 28-day intervals. After 3 cycles, bone marrow (BM) minimal residual disease (MRD) detection and efficacy evaluation (iwCLL2018 guidelines) are conducted. If BM MRD is negative (<10-4), patients will receive be treated with orelabrutinib plus obinutuzumab in 4-6 cycles; If BM MRD is positive (≥10-4), patients will receive the same regimen in 4-6 cycles as in previous 3 cycles. After 6 cycles of treatment, BM MRD detection and efficacy assessment will be conducted again. If BM MRD is negative (<10-4), orelabrutinib monotherapy will be administered in 7-12 cycles; If BM MRD is positive (≥10-4), treatment with orelabrutinib plus obinutuzumab will be administered in 7-12 cycles. After 12 cycles of treatment, BM MRD detection and efficacy evaluation will be performed. If BM MRD is negative (<10-4), orelabrutinib will be withdrawn and participants will turn to follow-up (efficacy assessment and MRD test will be performed according to the follow-up plan); if BM MRD is positive, treatment with orelabrutinib monotherapy will be administered in 13-24 cycles (continued even if BM MRD test was negative). After 24 cycles, if BM MRD is negative, the drug can be stopped and participants turn to follow-up. If BM MRD is positive, treatment can be continued until disease progression or be ceased by investigator due to no benefit from continued treatment, and BM MRD can be tested as planned. The trial is expected to end 36 months after enrollment of the last patient. If the subjects continue to require subsequent treatment with orelabrutinib, the sponsor will coordinate with the manufacturer and continue to provide the monotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 65 years old for both gender.
2. Patients have a confirmed diagnosis of CD20-positive chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) and meet criteria to initiate first-line treatment per International Workshop on CLL Working Group (IWCLL) 2018 guidelines
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. At least one measurable disease detected by enhanced computerized tomography (CT) or magnetic resonance imaging (MRI). At least one lymph node with the longest axis >=1.5cm and one measurable vertical dimension.
5. With life expectancy > 6 months.
6. Patients must meet the following laboratory examination criteria during 14 days before entry:

Serum bilirubin <1.5 Upper Limit of Normal (ULN), other than gilbert syndrome (defined as unconjugated bilirubin>80%); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 ULN.

Absolute neutrophil count (ANC)≥0.75×109/L and Platelets≥50×109/L (patients without exposure to G-CSF or blood transfusion within 7 days and no exposure to )

Exclusion Criteria:

1. Cumulative illness rating scale (CIRS) > 6.
2. Creatinine clearance rate (Ccr) <70 ml/min calculated by Cockcroft-Gault formula or by 24-hour urine analysis.
3. Patients diagnosed as other malignancy except lymphoma, except patients with curative intent and with no known active disease present for ≥ 5 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
4. Patients with known central nervous system involvement.
5. Patients with progressive multifocal leukoencephalopathy (PML).
6. Patients with history of Richter's Syndrome or suspected Richter's Syndrome.
7. Uncontrolled autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura, e.g. persistent decreasing hemoglobin or platelet count requiring steroid therapy 4 weeks before initiation of study.
8. Prior exposure to systemic therapy for CLL/SLL (except for incomplete treatment regimens fewer than 2 weeks such as antitumor steroid therapy).
9. Prior exposure to live vaccines, immunotherapy or other investigational therapeutic agent within 4 weeks prior to enrollment.
10. Requiring persistent steroid therapy for other non-antitumor purposes. Systemic steroid drug use within 7 days of first dose of study drug except regional use of steroid drug.
11. Uncontrolled or other serious cardiovascular disease, including:

    1. New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina, myocardial infarction, or clinically significant arrhythmia requiring medical intervention with a left ventricular ejection fraction (LVEF) <50% at screening 6 months prior to initial administration of the study drug;
    2. Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, rhythmogenesis right ventricular cardiomyopathy, restricted cardiomyopathy, unshaped cardiomyopathy);
    3. Clinically significant prolonged QTc interval, or QTc interval >470 ms in female and >450 ms in male at screening;
    4. Uncontrolled hypertension: on the basis of lifestyle improvement, blood pressure still fails to reach the standard after application of 2 or more kinds of reasonable, tolerable and full dose antihypertensive drugs (including diuretics), or 4 or more kinds of antihypertensive drugs until blood pressure can be effectively controlled.
12. Active bleeding within 2 months prior to screening, or taking anticoagulant/platelet drugs, or have a definite bleeding tendency in the investigator's opinion (e.g., esophageal varices with bleeding risk, local active ulcer lesions);
13. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
14. Clinically significant gastrointestinal abnormalities that may affect drug ingestion, transport, or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy.
15. Major surgery within 4 weeks of first dose of study drug. Diagnostic examination is not regarded as surgery and insertion of vascular access device excluded from the criteria.
16. Uncontrolled active systemic fungi, bacteria, virus (e.g. CMV DNA positive by PCR analysis) or other infections (defined as showing persistent symptoms of infection and no improvement although appropriate antibiotics or other treatment have been applied), or requiring intravenous (IV) antibiotics administration.
17. Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection (positive results from PCR analysis).
18. Known hypersensitivity to Orelabrutinib, Fludarabine, Cyclophosphamide or Obinutuzumab
19. Concurrent treatment with strong or moderate cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or inducers.
20. Any mental or cognitive impairment that may limit their understanding of informed consent and compliance with the study.
21. Pregnant and lactating women, or women of childbearing age who are unwilling to use contraception throughout the study period and within 18 months of the last administration of obinutuzumab or within 180 days of the last administration of any other study drug (women who were fertile must have a negative serological pregnancy test within 14 days prior to initiation of study) Male without surgically sterilized who are unwilling to use contraception throughout the study period and within 180 days of the last administration of the study drug.
22. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2025-02-22 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
BM undetectable MRD rate after 6 cycles | at the end of 6 cycles(each cycle is 28 days)
  Participants who achieve bone marrow (BM) undetectable Minimal Residue Disease (uMRD) after 6 cycles detecting by four-color flow cytometry with a detection level of 10-4.

SECONDARY OUTCOMES:
BM and PB undetectable MRD ratev after 3, 12, 24 cycles. | at the end of 3, 12, 24 cycles(each cycle is 28 days)
  participants who achieve BM uMRD (<10-4) on other important evaluation time-point (e.g. after 3, 12 and 24 cycles) except after 6 cycles. participants who achieve peripheral blood (PB) uMRD (<10-4) on important evaluation time-point.
Objective Response Rate (ORR) | at the end of 3, 6 cycles and up to approximately 3 years.(each cycle is 28 days)
  Response assessed after 3 and 6 cycles and up to approximately 3 years.
Complete Remission Rate (CRR) | at the end of 3, 6 cycles and up to approximately 3 years.(each cycle is 28 days)
  Response assessed after 3 and 6 cycles and up to approximately 3 years.
Duration of Response (DOR) | up to approximately 2, 3 years
  DOR is defined as duration in days from the data of initial documentation of objective response to the date of first documented evidence of progressive disease (PD) or death from any cause. Response and PD are defined according to iwCLL 2018 guidelines.
Progression Free Survival (PFS) | up to 3 years
  PFS is defined as duration from the date of enrollment to date of progressive disease, replase, or death from any cause, whichever occurs first. PD are defined according to iwCLL 2018 guidelines.
Overall Survival (OS) | up to 3 years
  OS is defined as the time from the date of enrollment to the date of the participant's death from any cause.
Incidence of adverse events (AEs) | through study completion, an average of 4 year"
  Treatment emergent adverse events (TEAE), severe adverse events (SAEs), adverse events of special interest (AESIs) and therapy-related AEs will be recorded and graded will be summarized by grade according to CTCAE (version 5.0).

OTHER OUTCOMES:
PB and BM Undetectable MRD rate by Next-generation Sequencing (NGS ) after 3, 6, 12 and 24 cycles. | at the end of 3, 6, 12 and 24 cycles(each cycle is 28 days)
  Participants who achieve BM and PB uMRD (<10-6) detected by NGS after 3 and 6 cycles. Participants who achieve BM uMRD (<10-6) detected by NGS after 12 and 24 cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, Phd, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Haematology, the First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjin, Jiangsu, China